CLINICAL TRIAL: NCT02902679
Title: An Open-label Study to Evaluate the Safety and Pharmacokinetics of BMS-986177 in Participants With End-stage Renal Dysfunction on Chronic Stable Hemodialysis Treatment
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of BMS-986177 in Participants With End-stage Renal Dysfunction on Chronic Stable Hemodialysis Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV010-012
Record Dates: First submitted 2016-08-24; First posted 2016-09-16 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Thrombosis; Factor XI; Renal Impairment; ESRD (End-Stage Renal Disease)
MeSH Terms: conditions — Thrombosis; Renal Insufficiency; Renal Insufficiency, Chronic | interventions — milvexian

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- End Stage Renal Disease Subjects (Experimental): Subjects given a single oral dose of BMS-986177 before (Period 1) and after (Period 2) a hemodialysis session
  Interventions: Drug: BMS-986177

INTERVENTIONS:
Drug: BMS-986177

SUMMARY:
An oral dose of BMS-986177 administered in End-stage Renal Dysfunction (ESRD) participants before and after a hemodialysis session to evaluate safety, tolerability, and pharmacokinetics in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Classified at screening as having ESRD requiring hemodialysis at least 3 times per week for 3 months.
* Clinical, ECG, and laboratory findings consistent with renal dysfunction
* BMI of 18.0 to 38.0 kg/m2 inclusive
* Subjects must receive unfractionated heparin during dialysis treatments and are able to withstand a decrease in their established heparin dose (75% of current dose)
* Women Not of child bearing potential (WNOCBP). Sexually active fertile men with partners who are WOCBP must use non-hormonal highly effective birth control

Exclusion Criteria:

* History of uncontrolled or unstable cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematopoietic, psychiatric, and/or neurological disease within 6 months of screening
* Evidence or history of coagulopathy, prolonged or unexplained clinically significant bleeding, or frequent unexplained bruising
* Current or recent (within 3 months of study drug administration) clinically significant gastrointestinal disease or gastrointestinal surgery that could interfere with absorption of study drug
* Any condition requiring anticoagulation such as, but not limited to, atrial fibrillation, mechanical prosthetic valve, deep venous thrombosis, or pulmonary embolism (other than heparin required during hemodialysis)
* Need for aspirin or need for P2Y12 antagonist therapy (for example clopidogrel, prasugrel, or ticagrelor)
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
To assess the Number of subjects with Adverse events (AEs). | Day -1 - day 3
To assess the Change from baseline in Physical examination parameters. | Day -1 - day 3
To assess the change from baseline in Electrocardiogram (ECG) assessment. | Day -1 - day 3
To assess the change from baseline in clinical laboratory values. | Day -1 - day 3
To assess the change from baseline in vital signs assessment. | Day -1 - day 3

SECONDARY OUTCOMES:
To assess the change from baseline in activated partial thromboplastin time (aPTT). | Day -1 - day 3
To assess the change from baseline in Factor XI clotting activity (FX1c ). | Day -1 - day 3

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States

REFERENCES:
- See also: BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/